CLINICAL TRIAL: NCT01487512
Title: A Single-Dose, Open-Label, Randomized, Crossover Dose Proportionality Study to Evaluate the Effect of Dose on the Pharmacokinetics of 8, 16, 32 and 64 mg OROS Hydromorphone Under Fasted Conditions in Healthy Adult Taiwanese Subjects
Brief Title: Effect of Dose on the Pharmacokinetics of OROS Hydromorphone Under Fasted Conditions in Healthy Taiwanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR017692; 42801PAI1010 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; Dose Proportionality; Pharmacokinetics; OROS Hydromorphone; Hydromorphone; Taiwan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence 1: Treatment A-D-B-C (Experimental): The study consists of 4 single-dose treatment periods. Successive drug administrations will be separated by a washout period of at least 7 and no more than 14 days.
  Interventions: Drug: Treatment A: Hydromorphone 8 mg; Drug: Treatment B: Hydromorphone 16 mg; Drug: Treatment C: Hydromorphone 32 mg; Drug: Treatment D: Hydromorphone 64 mg
- Sequence 2: Treatment B-A-C-D (Experimental): The study consists of 4 single-dose treatment periods. Successive drug administrations will be separated by a washout period of at least 7 and no more than 14 days.
  Interventions: Drug: Treatment A: Hydromorphone 8 mg; Drug: Treatment B: Hydromorphone 16 mg; Drug: Treatment C: Hydromorphone 32 mg; Drug: Treatment D: Hydromorphone 64 mg
- Sequence 3: Treatment C-B-D-A (Experimental): The study consists of 4 single-dose treatment periods. Successive drug administrations will be separated by a washout period of at least 7 and no more than 14 days.
  Interventions: Drug: Treatment A: Hydromorphone 8 mg; Drug: Treatment B: Hydromorphone 16 mg; Drug: Treatment C: Hydromorphone 32 mg; Drug: Treatment D: Hydromorphone 64 mg
- Sequence 4: Treatment D-C-A-B (Experimental): The study consists of 4 single-dose treatment periods. Successive drug administrations will be separated by a washout period of at least 7 and no more than 14 days.
  Interventions: Drug: Treatment A: Hydromorphone 8 mg; Drug: Treatment B: Hydromorphone 16 mg; Drug: Treatment C: Hydromorphone 32 mg; Drug: Treatment D: Hydromorphone 64 mg

INTERVENTIONS:
Drug: Treatment A: Hydromorphone 8 mg — type= exact number, unit= mg, number= 8, form= tablet, route= oral use. One tablet of Hydromorphone 8 mg in each of 4 treatment sequences.
Drug: Treatment B: Hydromorphone 16 mg — type= exact number, unit= mg, number= 16, form= tablet, route= oral use. One tablet of Hydromorphone 16 mg in each of 4 treatment sequences.
Drug: Treatment C: Hydromorphone 32 mg — type= exact number, unit= mg, number= 32, form= tablet, route= oral use. One tablet of Hydromorphone 32 mg in each of 4 treatment sequences.
Drug: Treatment D: Hydromorphone 64 mg — type= exact number, unit= mg, number= 64, form= tablet, route= oral use. One tablet of Hydromorphone 64 mg in each of 4 treatment sequences.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of OROS Hydromorphone in healthy adult Taiwanese participants after oral administration of 4 different dose strengths of 8, 16, 32 and 64 mg under fasted conditions.

DETAILED DESCRIPTION:
This is a single-center, randomized (study drug assigned by chance like flipping a coin), open-label (all people involved know the identity of the intervention), 4-way crossover (participants receive different interventions sequentially during the trial) study in healthy adult Taiwanese participants. All participants will be randomly assigned to 1 of the 4 different possible treatment sequences and will receive all treatments in the order specified by the randomization schedule. The study consists of a screening phase, an open-label treatment phase consisting of 4 single-dose treatment periods, and end-of-study or withdrawal assessments. During the open-label treatment periods, the participants will stay in the center until completion of the 72-hour pharmacokinetics [PK] (how the drug is absorbed in the body, distributed within the body, and how it is removed from the body over time) blood sample on Day 4. A 7- to 14-day washout period (period when receiving no treatment) will separate the open-label treatment periods. The safety and tolerability will be evaluated over the investigated dose range. The duration of participation in the study for an individual participant will be approximately 12 weeks.

ELIGIBILITY:
Inclusion Criteria: - Body mass index (BMI) between 18 and 25 kg/m², inclusive and a body weight of not less than 50 kg - Participants must utilize a medically acceptable method of contraception throughout the entire study period and for 1 month after the study is completed - Each participant will receive a naloxone challenge test for opioid dependency at screening. Only those participants who pass this challenge test will be allowed to continue in the study Exclusion Criteria: - History of or current clinically medical illness or any other condition that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results - Clinically significant abnormal values for hematology, clinical chemistry or urinalysis - Clinically significant abnormal physical examination, vital signs or 12 lead electrocardiogram (ECG) - Use of certain prescription or nonprescription medication, and consumption of products that may interfere with the study

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2011-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Plasma hydromorphone concentrations | 20 time points up to 72 hours post-dose
  Sequential blood samples are collected over 72 hours during each treatment period. The study has a total of four 5-day treatment periods. The treatment periods are separated by a 7- to 14-day washout period.

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Approximately 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Taipei, Taiwan